CLINICAL TRIAL: NCT01022047
Title: A Phase III, Non-inferiority, Open-label, Multicenter and Randomized Clinical Trial About the Treatment of Mild to Moderate Persistent Allergic Rhinitis in a Test Group Treated With Noex 32 mcg and a Reference Group Treated With Budecort Aqua® 32 mcg
Brief Title: Non-inferiority, Open-label, Multicenter and Randomized Clinical Trial About the Treatment of Mild to Moderate Persistent Allergic Rhinitis
Acronym: NOEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF096
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2010-12

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Noex (Experimental): The patients shall use the NOEX drug only once a day (one application in each nostril) during the 12 weeks of treatment
  Interventions: Drug: Noex
- Budecort Aqua (Active Comparator): The patients shall use the Budecort Aqua drug only once a day (one application in each nostril) during the 12 weeks of treatment.
  Interventions: Drug: Budecort Aqua

INTERVENTIONS:
Drug: Noex — The patients shall use the Noex drug only once a day (one application in each nostril) during the 12 weeks of treatment
  Arms: Noex
Drug: Budecort Aqua — The patients shall use the Budecort Aqua drug only once a day (one application in each nostril) during the 12 weeks of treatment.
  Arms: Budecort Aqua

SUMMARY:
To assess the efficacy of the study product Noex in the treatment of allergic rhinitis by means of the Nasal Index Score (NIS) after 4 weeks of treatment with the drug.

DETAILED DESCRIPTION:
Primary objective: To assess the efficacy of the study product Noex in the treatment of allergic rhinitis by means of the Nasal Index Score (NIS) after 4 weeks of treatment with the drug.

Secondary objectives: To determine the total NIS scale score after 12 weeks of treatment and the scores of the same scale individually for the symptoms of nasal obstruction, coryza, sneezing and nasal pruritus after 4 and 12 weeks of treatment, as well as to assess the safety of the study product according to the presence of adverse events.

Some eligibility criteria:

* NIS scale score > 4 points at the randomization visit
* Patients with persistent mild to moderate AR, according to the ARIA criteria with indication for use budesonide;

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form or - in case of patients younger than 18 years, the legal responsible must sign the consent;
* ≥ 12 years old;
* NIS scale score > 4 points at the randomization visit
* Patients with persistent mild to moderate AR, according to the ARIA criteria (see Appendix B), with indication for use budesonide;
* Positive skin test for at least one relevant airborne agent;
* AR symptoms for at least 2 years;
* May undergo a washout period of at least 2 weeks (without using any oral, nasal or inhalant corticosteroid agent; see 6.4).

Exclusion Criteria:

* Patients with persistent severe allergic rhinitis;
* Patients with severe co-morbidities (at the investigator's opinion);
* Patients with moderate to severe persistent asthma;
* Clinical history of infection of the airways 30 days before the study entry;
* Patients with structural changes causing nasal obstruction, such as pronounced nasal septum deviation, nasal polyps or any other type of nasal malformation;
* Pregnant women and patients planning to become pregnant during the study period or breastfeeding women;
* Patients in need of other drugs to treat the allergic rhinitis, such as anti-immunoglobulin E, allergen-specific immunotherapy, anti-leukotrienes, systemic vasoconstrictors, oral corticosteroids and other inhalant corticosteroids.

Patients using allergen-specific immunotherapy during the last year, as well as using anti-leukotrienes and anti-immunoglobulin E during the last month, or even patients using inhalant or oral corticosteroids after V0 will not be enrolled in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the efficiency of Noex | 5 months

SECONDARY OUTCOMES:
The secondary objectives and endpoints of the study are to evaluate the safety of Noex®, according to the frequency of the adverse events. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Morato, M.D., Principal Investigator — IMA Brasil - Instituto de Pesquisa Clínica e Medicina Avançada
Locations (1):
- IMA Brasil - Instituto de Pesquisa Clínica e Medicina Avançada, São Paulo, Brazil